CLINICAL TRIAL: NCT01913587
Title: Efficacy and Safety of Acupuncture on Spinal Compression Fracture in Patients Treated With Nerve Block
Brief Title: Efficacy Study of Acupuncture on Spinal Compression Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Jin Yong Jung, Department of anesthesiolgy, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIMI-13-01-21
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Spinal Compression Fracture
MeSH Terms: interventions — Acupuncture Therapy; Nerve Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture & Nerve block (Experimental): Acupuncture will be performed 3 times per week, total 9 sessions, during 3 weeks. Epidural nerve block and medial branch block will be performed once per week, total 3 sessions, during 3 weeks.
  Interventions: Device: Acupuncture; Procedure: Nerve block
- Nerve block (Active Comparator): Epidural nerve block and medial branch block will be performed once per week, total 3 sessions, during 3 weeks.
  Interventions: Procedure: Nerve block

INTERVENTIONS:
Device: Acupuncture — Acupuncture points are ST36, GB34 (bilateral), BL60 (bilateral), BL40 (bilateral), and 2 Back-su points (bilateral). Back-su points are selected as close as possible to pain region. Electroacupuncture will be performed at only 2 Back-su points (bilateral).
  Arms: Acupuncture & Nerve block
Procedure: Nerve block — Epidural nerve block uses the mixture (10ml) of dexamethasone (10 mg) and bupivacaine (10 mg) dissolved in saline solution. Medial branch block uses mepivacaine (10 mg).

SUMMARY:
This study is to investigate the effectiveness of acupuncture for alleviating pain from Spinal Compression Fracture in Patients Treated with Nerve Block.

DETAILED DESCRIPTION:
Spinal compression fracture is mainly caused by trauma, furthermore, in old age, osteoporosis increases the risk of spinal compression fracture. Nerve block is effective for the management of pain from inflammation or nerve root stimulation from spinal compression fracture. As one of alternative interventions, acupuncture is effective for controlling spinal compression fracture.

This study aims to investigate that combination with acupuncture and nerve block may relieve spinal compression fracture-related pain versus nerve block alone.

ELIGIBILITY:
Inclusion Criteria:

* Vertebral compression fracture by trauma or osteoporosis
* Minimum 15% height loss of vertebrae
* Patient diagnosed with x-ray or computed tomography (CT) or magnetic resonance image (MRI)
* Visual analogue scale (VAS) score of 5 or more
* Age over 50
* 2 weeks from onset or more
* Follow-up possible during the clinical trial
* Written informed consent voluntarily

Exclusion Criteria:

* Within 2 weeks from onset
* Pathological fracture due to malignancy/myeloma, osteomyelitis
* Major retropulsion of bony segments into the spinal canal
* Bone metabolic disease
* Significant renal or hepatic disease
* Hypersensitive reaction to acupuncture treatment
* Senile dementia, impaired cognitive function or other cerebral disease, severe psychiatric or psychological disorders
* Alcohol/drug abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | Change from baseline to 5 weeks
  The patients will be required to document 100mm pain VAS, where '0' represents 'no pain' and '100', 'unbearable pain'. The change of pain will be reported by comparing the mean VAS before treatment, after 3 week, and 5 week (2 weeks follow-up).

SECONDARY OUTCOMES:
Short form McGill pain questionnaire | Change from baseline to 5 weeks
  Evaluation will performed before treatment, after 3 week, and 5 week (2 weeks follow-up).
Oswestry Disability Index (ODI) | Change from baseline to 5 weeks
  Evaluation will be performed before treatment, after 3 week, and 5 week (2 weeks follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Chul Seo, KMD, Ph.D, Principal Investigator — Comprehensive and Intergrative Medicine Institute; Min-Ah Gwak, KMD, Ph.D, Principal Investigator — Daegu Oriental Hospital of Daegu Haany University; Seong-Hoon Park, KMD, Principal Investigator — Comprehensive and Integrative Medicine Insitute
Locations (1):
- Daegu Catholic University Medical Center, Daegu, Kyungsangbukdo, South Korea